CLINICAL TRIAL: NCT02226874
Title: A Comparison of Two Dose Assessment Methods for Exposures to Nuclear Detonation Radiation
Brief Title: Comparison of Two Dose Assessment Methods for Exposures to Nuclear Detonation Radiation
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999914170; 14-C-N170
Record Dates: First submitted 2014-08-26; First posted 2014-08-27 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2019-04-24

CONDITIONS: Radiation Exposure
Keywords: Dose Estimation; Dose Reconstruction; Methods; Fallout; Radiation Exposure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

SUMMARY:
Background:

- The National Cancer Institute was funded to study how much radiation U.S. veterans who served in the 1950s were exposed to. Researchers want to estimate how much radiation these veterans received. They will use two methods and compare them. One is to interview the veterans and study their military records. The other is to take blood samples and look for certain types of changes in the blood cells. Being exposed to some kinds of radiation is known to cause changes in blood cells. The amount of changes to these cells tells scientists about how much radiation was received.

Objectives:

- To better understand how to measure how much radiation a person has received.

Eligibility:

* Veterans who were exposed to radiation at a specific site in the Pacific in 1954 or other sites in the 1950s.
* Veterans close in age to the first group, who have low levels of exposure to radiation.
* Men about 25 years old with no exposure to radiation.

Design:

* Participants will have 1 visit, in their home.
* All participants will have blood drawn. This will take 10 minutes.
* The exposed veterans will be interviewed. They will answer questions about the nuclear events they experienced. This will take up to 40 minutes.
* For the exposed veterans, researchers will look at their military records, if they can. They will estimate how much radiation the veteran received.

DETAILED DESCRIPTION:
Understanding the potential consequences of exposures from nuclear detonations is a current national security concern. In the event of a nuclear detonation, an important priority for the scientific and national security community is to be able to estimate exposure to the general population for medical triage, treatment, follow-up and risk projection for public health purposes. The only available comprehensive exposure estimates for persons exposed to nuclear detonation radiation are from studies of wartime atomic bomb survivors. There is an urgent need to evaluate exposure assessment methods in other populations and to determine how well each works and the obstacles involved in the application of each.

In the absence of other studies of exposures to nuclear detonation radiation, the Atomic Veterans Epidemiologic Study (AVES)1, a large ongoing study of atomic veterans of 115,000 atomic veterans who participated in aboveground nuclear weapon tests during 1945-1962 provides a unique opportunity to evaluate the lasting biological effects of radiations received during nuclear detonations. That study has the means for identifying veterans who received the highest exposures as well as control subjects with minimal to no exposure. An overview of the AVES can be found at http://www.vbdr.org/meetings/2013/Presentations/02_Dr_Boice.pdf.

We propose to conduct a small methodologic investigation with the following objective: evaluate the level of agreement between radiation exposure estimates from the generally simple and inexpensive assessment strategy of model-based dose reconstruction with the only well-established long-term biologically-based dose estimation technique - quantification of chromosome aberration frequency. In this study, the dose reconstruction would include individual interview data.

The study would be conducted using a group of U.S. veterans exposed to nuclear detonation radiation during the 1950s and 1960s. While there are many thousands of veterans still alive today who participated in nuclear testing-related activities, only 16 have been identified that are still living and that have estimated exposures of sufficient magnitude for the chromosome aberration frequency assay to be successful. These particular veterans were exposed on Rongerik Atoll in the Pacific in 1954 and at the Nevada Test Site in 1951-1952. The dose estimates will also be compared against individual records of exposure obtained from radiation film-badges, when available. All the persons to be studied are part of the study cohort in the AVES study.

The primary purpose of evaluating the model-based dose reconstruction with the dose estimates based on chromosome aberration frequency will be to assess the presence of any substantial differences (either systematic or random) in doses now being estimated via model-based dose reconstruction in the AVES. Because the chromosome aberration frequency assay is difficult, expensive and somewhat invasive (requiring a blood sample), it is not practical in a study of many thousands of subjects as in the AVES. Determination that the model-based dose estimations are not systematically different from FISH-estimated doses is of substantial value to the AVES. To a limited degree, i.e., within the constraints of the small sample size, the study may be indicative of the potential for model-based dose estimates to be relied upon if mass exposures were to take place from a nuclear detonation.

It is noteworthy that the collection of samples and data to evaluate doses in this study will take advantage of a one-of-a-kind situation to obtain exposure-related data from a unique (and rapidly dwindling) population living persons exposed to atomic weapons detonation radiation a situation that cannot be repeated except under wartime or actual national threat situations.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

EXPOSED VETERANS. Subjects for this investigation are required to have received, according to military records, whole-body radiation doses in excess of 0.25 Sv to ensure adequate detection of the radiation exposure by the FISH method. The recorded doses are crude dose estimates, often based on group radiation monitoring rather than on individual data, however, they are the only information available, upon which to select the study subjects that meet our criteria.

To date, 16 exposed veterans that meet this requirement have been identified by the AVES through accessing databases of the NTPRP constructed by the Dept. of Defense.

Ages: 80 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-08-26; Primary Completion 2016-05-31 (Actual); Study Completion 2016-05-31 (Actual)

PRIMARY OUTCOMES:
Dosimetry data | September 2014 - December 2016
  Comparing dosimetry data between cases and controls

CONTACTS AND LOCATIONS:
Overall Officials: Steven L Simon, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Colorado State University, Fort Collins, Colorado, United States

REFERENCES:
- [Background] Edwards AA, Szluinska M, Lloyd DC. Reconstruction of doses from ionizing radiation using fluorescence in situ hybridization techniques. Br J Radiol. 2007 Sep;80 Spec No 1:S63-7. doi: 10.1259/bjr/24766640. PMID 17704328
- [Background] Hande MP, Azizova TV, Geard CR, Burak LE, Mitchell CR, Khokhryakov VF, Vasilenko EK, Brenner DJ. Past exposure to densely ionizing radiation leaves a unique permanent signature in the genome. Am J Hum Genet. 2003 May;72(5):1162-70. doi: 10.1086/375041. Epub 2003 Apr 4. PMID 12679897
- [Background] Sigurdson AJ, Ha M, Hauptmann M, Bhatti P, Sram RJ, Beskid O, Tawn EJ, Whitehouse CA, Lindholm C, Nakano M, Kodama Y, Nakamura N, Vorobtsova I, Oestreicher U, Stephan G, Yong LC, Bauchinger M, Schmid E, Chung HW, Darroudi F, Roy L, Voisin P, Barquinero JF, Livingston G, Blakey D, Hayata I, Zhang W, Wang C, Bennett LM, Littlefield LG, Edwards AA, Kleinerman RA, Tucker JD. International study of factors affecting human chromosome translocations. Mutat Res. 2008 Apr 30;652(2):112-21. doi: 10.1016/j.mrgentox.2008.01.005. Epub 2008 Feb 2. PMID 18337160